CLINICAL TRIAL: NCT02822287
Title: An Open Label Study to Assess the Warming Sensation, Acceptability and Local Oral Tolerability of NCH-GSK Acetylcysteine 2% Oral Solution, Given as a Single Dose in Subjects Suffering From Productive Cough Due to Upper Respiratory Tract Infection
Brief Title: Warming Sensation and Tolerability Study of Acetylcysteine 2% Oral Solution for Productive Cough
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205034
Record Dates: First submitted 2016-02-11; First posted 2016-07-04 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-09

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — N-monoacetylcystine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2% Acetylcystine Solution (Experimental): Participants will be orally administered with the clear oral solution containing 2% acetylcysteine (g/mL) in a 100 mL amber glass bottle over 1 minute or less using an oral syringe.
  Interventions: Drug: Acetylcystine

INTERVENTIONS:
Drug: Acetylcystine — Clear oral solution containing 2% acetylcysteine (g/mL) in a 100 mL amber glass bottle.

SUMMARY:
This is a 1-treatment arm, open label design. This 1-day study includes a screening on day of attendance at clinic, followed by a washout period of 30 minutes to 8 hours (if participants are eligible for dosing the same day). The study also includes a supervised dosing with 10 mL oral solution and a 1 hour in-clinic evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must give written informed consent before any assessment is performed. In the case of adolescents Informed Consent must be signed by one or both parents or legal guardian as per local regulations and an Informed Assent must be signed by the participant.
* Must be males or females ≥ 12 years.
* Willingness and ability to communicate, to comply with all study requirements and to complete the study.
* Productive cough of less than 7 days duration, rated based on interview with the participant as mild to moderate severity on a four- point ordinal scale (not present, mild, moderate, severe) due to upper respiratory tract infection.

Exclusion Criteria:

* Use of other investigational drugs before enrollment, or within 30 days or 5 half-lives before enrollment, whichever is longer.
* Pre-dose productive cough or sore throat rated as severe on a four-point ordinal scale (not present, mild, moderate, severe) based on interview with the participant.
* Pre-dose temperature equal or above 39.4°C at screening measured by oral thermometer.
* History of hypersensitivity to any of the study drugs and the listed excipients or to drugs of similar chemical classes.
* Pregnant , nursing (lactating women) or women with child bearing potential UNLESS they are using effective methods of contraception.
* Use of any medication for sore throat containing a local anaesthetic, methanol or any topical products containing menthol, peppermint, spearmint or within the 6 hours prior to dosing.
* Use of any paracetamol, non-steroidal anti-inflammatory drug (NSAID) or any oral/nasal decongestant within 6 hours prior to dosing.
* Use of substances of abuse, herbal medications, or antihistamines within 48 hours of dosing.
* Hepatic or severe renal impairment, hypertension, hyperthyroidism, diabetes, or heart disease.
* Drinking of tea, coffee or other caffeinated beverages 1 hour prior to dosing.
* Drinking of any hot beverages 1 hour prior to dosing.
* Participant is a current smoker of ≥10 cigarettes per day (or reports equivalent smoking habits using other tobacco products) or smoked or chewed tobacco products within 12 hours before dosing.
* Participant is taking nitroglycerin and nitrate drug treatments.
* Participants who took antibiotic treatments such as semisynthetic penicillins, tetracyclines, cephalosporins and aminoglycosides within 2 hours of dosing. Amoxicillin, doxycycline, erythromycin, thiamphenicol and cefuroxime are allowed without this restriction.
* Participants with gastroduodenal (peptic) ulcers, asthma.
* Participants with intolerance to histamines.
* Participants who have used antitussives (e.g., dextromethorphan, codeine), anticholinergic drugs (atropine-like) within the past 24 hours.
* Participants who have taken heavy metal salts such as calcium, gold and iron within 2 hours of enrollment.
* A history of alcohol abuse or an admission by the participant that they regularly consume alcohol in excess of the recommended weekly limits of 21 units for females and 28 units for males.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Erfurt, Thuringia, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited at 1 center in Germany
Pre-assignment Details: A total of 58 potential participants were screened and 57 participants were included in the study. All 57 participants received the investigational product.
Groups:
- 2% Acetylcystine Solution: Participants received a single dose of 200 mg (10 mL) of Acetylcysteine 2% oral solution.
Period: Overall Study
Arm/Group | 2% Acetylcystine Solution
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population was the primary population. The Safety Population was defined as all treated subjects, i.e., all subjects who received any dose of study drug.
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (13.88)
Gender [Count of Participants; unit: Participants]
  Female | 33
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Onset of Warming Sensation
Description: Onset and duration of action of warming sensation was measured by two stop watches started when the participants took the oral solution. First watch was stopped at the start of warming sensation and the second watch was stopped at the end. If onset had not occurred by 10 minutes then time to onset was censored at 10 minutes. 53 of the 57 participants had onset within 10 minutes after dosing.
Time Frame: 10 minutes post-dose
Population: The Safety Population was defined as all treated subjects, i.e., all subjects who received any dose of study drug. The Safety Population was the primary population for both the primary and secondary endpoint analyses and the safety analysis.
Measure: Median (Full Range); unit: Minutes
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 57
Minutes | 0.233 [0.067 to 10.00]

2. Primary Outcome: Duration of Warming Sensation
Description: Duration of action of warming sensation was measured by two stop watches started when the participants took the oral solution. First watch was stopped at the start of warming sensation and the second watch was stopped at the end. If onset of warming sensation occurred within 10 minutes of dosing but had not ended by the end of 10 minutes following dosing, then the duration was censored at 10 minutes minus the time to onset
Time Frame: 10 minutes post-dose
Population: The safety Population was defined as all treated subjects, i.e., all subjects who received any dose of study drug. The Safety Population was the primary population for both the primary and secondary endpoint and safety analysis. Of the 57 subjects in the Safety Population, 53 reported an onset of a warming sensation within10 minutes after dosing.
Measure: Median (Full Range); unit: Minutes
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 53
Minutes | 2.833 [0.150 to 9.783]

3. Primary Outcome: Warming Sensation Intensity at Pre-Dose and 60 Sec (Seconds) Post-Dose
Description: Warming Sensation Intensity was measured on 100 mm visual analogue scale (VAS), marked as "no warming sensation" on the left hand side (= 0 mm) and "strongest possible warming sensation" at the right hand side (=100 mm) at pre-dose.
Time Frame: Pre-dose and 60 sec post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 57
Millimeters (mm)
  Pre-dose | 6.8 (8.69)
  Post-dose (Observed) | 36.1 (26.93)
  Post-dose (Change) | 29.2 (27.84)

4. Secondary Outcome: Number of Participants With Acceptability of Warming Sensation
Description: Acceptability of strength of warming sensation was measured by a scale: 5= Much too strong; 4=Too strong (too warming); 3= Just about right (pleasant warming); 2= Too weak (not warming enough); 1= Much too weak
Time Frame: 10 minutes post-dose
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 57
Number of Participants
  Much too strong | 0
  Too strong | 2
  Just about right | 30
  Too Weak | 16
  Much too weak | 9

5. Secondary Outcome: Number of Participants With Overall Opinion of Warming Sensation
Description: Overall opinion of warming sensation was measured by scale: 9= Like extremely; 8= Like very much; 7= Like moderately; 6= Like slightly; 5= Neither like nor dislike; 4= Dislike slightly; 3= Dislike moderately; 2= Dislike very much; 1= Dislike extremely
Time Frame: 10 minutes post-dose
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 57
Number of Participants
  Like extremely | 1
  Like very Much | 21
  Like moderately | 11
  Like slightly | 7
  Neither Like nor Dislike | 10
  Dislike slightly | 3
  Dislike Moderately | 1
  Dislike Very Much | 3
  Dislike extremely | 0

6. Secondary Outcome: Number of Participants With Overall Opinion of Oral Solution
Description: Overall opinion of oral solution was measured by scale: 4 = Excellent; 3 = Good; 2 = Fair; 1 = Poor; 0 = Unacceptable.
Time Frame: 1 hour post-dose
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 57
Number of Participants
  Excellent | 2
  Good | 21
  Fair | 29
  Poor | 5
  Unacceptable | 0

7. Secondary Outcome: Local Oral Tolerability
Description: Local oral tolerability was assessed by performing oropharyngeal examination as follows: Results of oropharyngeal examination (Normal and abnormal); If abnormal, any signs of lesion on oral mucosa or irritation of oral mucosa.
Time Frame: Day 1 (at screening and end of study)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 2% Acetylcystine Solution
Number analyzed (Participants) | 57
Participants
  Oropharyngeal examination at screening (Normal) | 52
  Oropharyngeal examination at study end (Normal) | 52
  Oropharyngeal examination at screening (Abnormal) | 5
  Oropharyngeal examination at study end (Abnormal) | 5
  Abnormal (lesions on oral mucosa) | 0
  Abnormal (No lesions on oral mucosa) | 5
  Abnormal (Irritation of oral Mucosa) | 0
  Abnormal (No irritation of oral Mucosa) | 5

ADVERSE EVENTS:
Arm/Group | 2% Acetylcystine Solution
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.